CLINICAL TRIAL: NCT05492266
Title: Expiratory Muscle Strength Training as a Non-surgical Option for Velopharyngeal Dysfunction: A Randomized-controlled Trial
Brief Title: Expiratory Muscle Strength Training for Hypernasal Speech in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noel Jabbour (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Noel Jabbour, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120032; 5R21DC017553-03 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Velopharyngeal Insufficiency; Velopharyngeal Incompetence Due to Cleft Palate; Inadequate Velopharyngeal Closure; Palatopharyngeal Incompetence; Hypernasality
Keywords: Cleft Palate; Speech Intelligibility
MeSH Terms: conditions — Velopharyngeal Insufficiency; Cleft Palate; Speech Intelligibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Expiratory Muscle Strength Training + No Maintenance Training (Experimental): These participants were initially randomized to complete 6-8 weeks of exercises with EMST-150. They had improvement in their CAPS-A hypernasality rating of 1 point or more and were randomized to complete 6 months of no maintenance training.
  Interventions: Device: Expiratory Muscle Strength Training
- No Exercises (No Intervention): These participants were initially randomized to 6-8 weeks of no exercises. They ended active study participation after the initial 6-8 weeks of no exercises. They were not eligible to be randomized to maintenance training or no maintenance training.
- Expiratory Muscle Strength Training + Maintenance Training (Experimental): These participants were initially randomized to complete 6-8 weeks of exercises with EMST-150. They had improvement in their CAPS-A hypernasality rating of 1 point or more and were randomized to complete 6 months of maintenance training.
  Interventions: Device: Expiratory Muscle Strength Training; Device: Maintenance Training
- Expiratory Muscle Strength Training (Experimental): These participants were initially randomized to complete 6-8 weeks of exercises with EMST-150. They did not have improvement in their CAPS-A hypernasality rating of 1 point or more and ended active study participation after the initial 6-8 weeks of exercises.
  Interventions: Device: Expiratory Muscle Strength Training

INTERVENTIONS:
Device: Expiratory Muscle Strength Training — At visit 1, participants will be block randomized based on PWSS score (5-6 or 7+) to Expiratory Muscle Strength Training (EMST) for 6 to 8 weeks or no exercises. Participants in the EMST-150 group will perform 5 sets of 5 resistive expirations once a day with a 10-15 second rest between each repetition and a 1-2 minute rest between each set of 5 repetitions.
  Other Names: EMST-150
  Arms: Expiratory Muscle Strength Training; Expiratory Muscle Strength Training + Maintenance Training; Expiratory Muscle Strength Training + No Maintenance Training
Device: Maintenance Training — At visit 2, participants with improved (decreased) CAPS-A hypernasality rating of 1 or more points, for whom the family and/or surgeon is not currently considering surgical intervention for VPI, will be further randomized to continue "maintenance" EMST exercises or no exercises for 6 months. Participants in the "maintenance" group will complete 3-5 sessions exercise sessions each week (rather than daily training), with 2 sets of 5 resistive expirations (rather than 5 sets)
  Arms: Expiratory Muscle Strength Training + Maintenance Training

SUMMARY:
When the soft palate does not move enough because of a cleft palate or for unknown reasons, this can lead to a speech difference called velopharyngeal insufficiency. The purpose of this research study is to test if soft palate exercises using a hand help breathing device will help improve the ability of the soft palate to close the area between the throat and nose and help improve speech.

DETAILED DESCRIPTION:
The objective of this study is to examine the feasibility and efficacy of expiratory muscle strength training to improve velopharyngeal closure in patients with velopharyngeal dysfunction and nasal air emissions. A randomized, controlled trial will be conducted at a cleft craniofacial center at a tertiary children's hospital. Patients will be block randomized based on Pittsburgh Weighted Speech Scale (PWSS) score (5-6 or 7+) to Expiratory Muscle Strength Training for 6 to 8 weeks or no exercises. Patients with reductions in nasal resonance during this time will be further randomized to EMST maintenance training for 6 months or no exercises.

ELIGIBILITY:
Inclusion Criteria:

* Pittsburgh weighted speech scores of 5 or greater
* Ages 5-17 years

Exclusion Criteria:

* CAPS-A-AM hypernasality score <2
* Previous speech surgery (e.g. palatoplasty or pharyngeal flap)
* Speech surgery scheduled within the next 56 days
* Unable or unwilling to perform the tests and exercises outlined in the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in nasalance scores after 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Percent change in nasalance measured during nasometry
Change in perceptual speech symptoms of velopharyngeal dysfunction following 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Perceptual symptoms of velopharyngeal incompetence measured using the CAPS-A-AM hypernasality score, on a scale of 0-4. 0 indicates nasality that is normal for the region, 1 (borderline/minimal) suggests a minimal or inconsistent increase in nasal resonance, 2 (mild) implies hypernasality that is evident on vowels with a high tongue posture, 3 (moderate) indicates hypernasality that is perceived across all vowels, and 4 (severe) signifies that hypernasality is evident in voiced consonants and all vowels.
Change in oral pressure following 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Percent change in oral pressure achieved when blowing through the EMST-150
Change in velopharyngeal flutter following 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Change in percentage of participants with oscillating oral pressure when blowing through the EMST-150
Change in oral pressure decay following 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Ratio of the magnitude of oral pressure decay when blowing through the EMST-150

SECONDARY OUTCOMES:
Change in VELO questionnaire scores following 6-8 weeks of exercises compared with baseline | Baseline and 6-8 weeks
  Percent change in Velopharyngeal Insufficiency (VPI) Effects on Life Outcomes (VELO) scores. Scores range from 0 - 100, with 100 representing the highest QOL
Resolution of type B tympanogram following 6-8 weeks of exercises compared with baseline. | Baseline and 6-8 weeks
  Percentage of participants with a change in tympanogram type from type B (flat) to type A (normal middle ear function).
Resolution of type C tympanogram following 6-8 weeks of exercises compared with baseline. | Baseline and 6-8 weeks
  Percentage of participants with a change in tympanogram type from type C (negative pressure) to type A (normal middle ear function).
Resolution of effusion following 6-8 weeks of exercises compared with baseline. | Baseline and 6-8 weeks
  Percentage of participants with resolution of middle ear effusion based on otoscopy.
Resolution of retraction following 6-8 weeks of exercises compared with baseline. | Baseline and 6-8 weeks
  Percentage of participants with resolution of tympanic membrane retraction based on otoscopy

OTHER OUTCOMES:
Change in nasalance scores after 6 months of maintenance exercises compared with after the initial 6-8 weeks of exercises | 6-8 weeks and 8 months
  Percent change in nasalance measured during nasometry
Change in perceptual speech symptoms of velopharyngeal dysfunction after 6 months of maintenance exercises compared with after the initial 6-8 weeks of exercises | 6-8 weeks and 8 months
  Perceptual symptoms of velopharyngeal incompetence measured using the CAPS-A-AM hypernasality score, on a scale of 0-4. 0 indicates nasality that is normal for the region, 1 (borderline/minimal) suggests a minimal or inconsistent increase in nasal resonance, 2 (mild) implies hypernasality that is evident on vowels with a high tongue posture, 3 (moderate) indicates hypernasality that is perceived across all vowels, and 4 (severe) signifies that hypernasality is evident in voiced consonants and all vowels.
Change in oral pressure after 6 months of maintenance exercises compared with after the initial 6-8 weeks of exercises | 6-8 weeks and 8 months
  Percent change in pressure achieved when blowing through the EMST-150
Change in velopharyngeal flutter after 6 months of maintenance exercises compared with after the initial 6-8 weeks of exercises | 6-8 weeks and 8 months
  Change in percentage of participants with oscillating oral pressure when blowing through the EMST-150
Change in oral pressure decay after 6 months of maintenance exercises compared with after the initial 6-8 weeks of exercises | 6-8 weeks and 8 months
  Ratio of the magnitude of oral pressure decay when blowing through the EMST-150
Prevalence of surgical intervention | 1 year
  Percentage of patients undergoing surgical intervention for speech symptoms within the 1 year following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Noel Jabbour, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in a publication may be shared, after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication of summary data. Ending 5 years after publication.
Access Criteria: IPD will be shared with researchers who provide a methodologically sound proposal. IPD to be shared will include that necessary to achieve the aims in the approved proposal. Proposals should be directed to shafferad@upmc.edu. To gain access, data requestors will need to sign data access agreement.